CLINICAL TRIAL: NCT02324907
Title: The Use of a Dynamic Compression Intramedullary Nail for Tibiotalocalcaneal Arthrodesis
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: MedShape, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00055335
Record Dates: First submitted 2014-12-16; First posted 2014-12-24 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2022-03

CONDITIONS: Ankle Arthritis
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tibiotalocalcaneal arthrodesis with DynaNail: Procedure/Surgery: Tibiotalocalcaneal arthrodesis with a novel dynamic compression intramedullary nail
  Interventions: Device: Procedure/Surgery

INTERVENTIONS:
Device: Procedure/Surgery — Tibiotalocalcaneal (TTC) arthrodesis with a novel dynamic compression intramedullary nail. The assignment of the device is at the discretion of the standard of care provider, not the study investigator.

SUMMARY:
The purpose of this study is to determine the clinical efficacy of a novel dynamic compression intramedullary nail for tibiotalocalcaneal (TTC) arthrodesis.

DETAILED DESCRIPTION:
This proposal is a collaborative effort of MedShape. This is a prospective investigation to assess the clinical outcomes of patients with a tibiotalocalcaneal arthrodesis with the Dynamic Compression Intramedullary Nail (DynaNail). We are planning on enrolling 30 patients. The assignment of the device is at the discretion of the standard of care provider, not the study investigator.

Patients with end-stage tibiotalar (ankle) and talocalcaneal (subtalar) joint arthritis from any etiology will be asked to enroll in the study. After informed consent, the patients will be asked to complete the following patient reported outcomes questionnaires (standard of care for all patients in the Foot and Ankle section): 100mm VAS for pain, Short form-36 (SF-36), and the Foot and Ankle Ability Measure (FAAM). After informed consent, they will then be scheduled for surgery in a routine fashion. REDCap database will be used to allow on-line data entry.

The following surgical procedure steps and follow-ups are standard of care at Duke University. The surgical procedure will involve both tibiotalar and talocalcaneal joint preparation through any approach (lateral, posterior, anterior with sinus tarsi). The use of supplemental bone graft is at the discretion of the treating surgeon but must be documented. The MedShape DynaNail will then be inserted according to the manufacturer's technique. The patient will be placed in a short leg splint and kept non-weight bearing. The patient will be discharged from the hospital when medically ready and follow-up in two weeks.

At two weeks, the patient will return to clinic for a standard of care visit and their splint will be removed. A non-weight bearing lateral radiograph of the hind foot will be taken to assess the amount of travel of the compressive element. This radiograph is not standard of care. The patient will be placed in a non-weight bearing cast. The patient will then be asked to return in two weeks (4 weeks post-operatively). This visit is not standard of care. At this time another non-weight bearing lateral radiograph will be taken to assess the amount of travel of the compressive element. The patient will be asked to return at 6 weeks, 3 months, 6 months, 12 months, and 24 months after surgery as is standard of care for this surgery. At 3 months, a CT scan will be obtained to assess healing. This is standard of care at Duke University. At each of these time-points, the same patient specific outcome questionnaires will be administered. For any non- standard of care radiographs patients will be asked to take a urine pregnancy test prior to any radiographs being taken.

Patients will be identified in the clinic by an attending orthopaedic foot and ankle surgeon or his physician assistant based on clinical exam and radiographic findings. Inclusion criteria include anyone over age 18 who has ankle and subtalar arthritis and has failed nonoperative management. Typically, these patients have multiple medical comorbidities and therefore the only exclusion criteria will be patients who are not healthy enough to undergo surgery. Patients of all racial, religious, and cultural backgrounds will be included in this study. Approximately 30 patients will be recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Ankle and Subtalar arthritis
* Failed non-operative management

Exclusion Criteria:

* Patients who do not meet the minimum age of 18 years.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified in the clinic by an attending orthopaedic foot and ankle surgeon or his physician assistant based on clinical exam and radiographic findings. Inclusion criteria include anyone over age 18 who has ankle and subtalar arthritis and has failed nonoperative management. Typically, these patients have multiple medical comorbidities and therefore the only exclusion criteria will be patients who are not healthy enough to undergo surgery. Patients of all racial, religious, and cultural backgrounds will be included in this study. Approximately 30 patients will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Change in Pain Assessment | Pre-operative up to 2 years post surgery
  Visual Analog Scale (VAS)
Change in Functional Assessment | Pre-operative up to 2 years post surgery
  Short Form 36 (SF-36)
Change in Functional Assessment | Pre-operative up to 2 years post surgery
  Foot and Ankle Ability Measure (FAAM)
Fusion, as measured by radiograph and CT scan | Pre-operative up to 2 years post surgery
  radiographs taken Pre-operatively, 2 weeks, 4 weeks, 6 weeks, 3 Months, 6 Months, 12 Months and 24 Months. A CT scan will be done standard of care at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Easley, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No